CLINICAL TRIAL: NCT00000626
Title: Phase II Study of Filgrastim (G-CSF) Plus ABVD in the Treatment of HIV-Associated Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 149; 11124 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hodgkin's Disease
Keywords: Granulocyte Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; Antineoplastic Agents, Combined; AIDS-Related Complex; Hodgkin Disease; ABVD protocol
MeSH Terms: conditions — HIV Infections; Hodgkin Disease; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Vinblastine; Dacarbazine; Filgrastim; Bleomycin; Doxorubicin

INTERVENTIONS:
Drug: Vinblastine sulfate
Drug: Dacarbazine
Drug: Filgrastim
Drug: Bleomycin sulfate
Drug: Doxorubicin hydrochloride

SUMMARY:
Primary: To assess the toxicity of chemotherapy with ABVD (doxorubicin / bleomycin / vinblastine / dacarbazine) when given with filgrastim ( granulocyte colony-stimulating factor; G-CSF ) in patients with underlying HIV infection and Hodgkin's disease; to observe the efficacy of ABVD and G-CSF in reducing tumor burden in HIV-infected patients with Hodgkin's disease.

Secondary: To determine the durability of tumor response to ABVD plus G-CSF over the 2-year study period; to observe the incidence of bacterial and opportunistic infections in HIV-infected patients with Hodgkin's disease receiving this regimen; to document quality of life of patients receiving this regimen.

Addition of granulocyte colony-stimulating factor may prevent neutropenia caused by chemotherapy, allowing more timely administration of chemotherapy and improved response.

DETAILED DESCRIPTION:
Addition of granulocyte colony-stimulating factor may prevent neutropenia caused by chemotherapy, allowing more timely administration of chemotherapy and improved response.

Study drugs are administered in 28-day cycles to twenty-seven HIV-infected patients with Hodgkin's disease. ABVD (doxorubicin / bleomycin / vinblastine / dacarbazine) is administered on days 1 and 15 of each cycle, and G-CSF is given on days 2 through 14 and 16 through 28 of each cycle. All patients receive four cycles of treatment and are then restaged. Patients with a complete response (CR) following the initial four cycles receive two additional cycles of ABVD / G-CSF. Patients with a partial response following the initial four cycles receive two additional cycles of ABVD / G-CSF and are again restaged; those who have achieved a CR at that point then receive two more cycles, while those without CR discontinue study therapy. Patients with disease progression following the initial four cycles of therapy discontinue treatment on the study. Concomitant PCP prophylaxis is administered.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* PCP prophylaxis consisting of Bactrim, aerosolized pentamidine, or dapsone.

Recommended:

* Antiemetic therapy within 30 minutes of chemotherapy.

Allowed:

* Antiretroviral medication after two cycles of chemotherapy, provided the patient has not experienced grade 3 neutropenia while on chemotherapy or on previous antiretroviral therapy.
* Acetaminophen and/or nonsteroidal anti-inflammatory agents.
* Bone marrow-suppressive agents, such as ganciclovir, Fansidar, Bactrim, and dapsone.
* Maintenance therapy for chronic opportunistic infection.

Concurrent Treatment:

Allowed:

* Cranial irradiation (2400 rads) for patients with CNS involvement.

Patients must have:

* Documented HIV infection or diagnosis of AIDS.
* Hodgkin's disease.
* Consent of parent or guardian and have care directly supervised by a pediatric oncologist if under 18 years of age.

Prior Medication:

Allowed:

* Maintenance therapy for opportunistic infections.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Second primary cancer other than Kaposi's sarcoma that does not require systemic therapy, nonmelanomatous skin cancer, Bowen's disease, or carcinoma in situ of the cervix.
* Acute, active bacterial or opportunistic infection requiring ongoing therapy if such therapy has been initiated within the past 2 weeks.
* Known hypersensitivity (e.g., anaphylactoid reaction, bronchospasm) to E. coli-derived proteins.

Prior Medication:

Excluded:

* Prior chemotherapy for Hodgkin's disease.
* Antiretroviral therapy within 2 weeks prior to study entry.

Prior Treatment:

Excluded:

* Prior radiotherapy for Hodgkin's disease.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27
Dates: Study Completion 1999-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Levine A, Study Chair
Locations (8):
- United States (8):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio

REFERENCES:
- [Background] Levine AM, Li P, Cheung T, Tulpule A, Von Roenn J, Nathwani BN, Ratner L. Chemotherapy consisting of doxorubicin, bleomycin, vinblastine, and dacarbazine with granulocyte-colony-stimulating factor in HIV-infected patients with newly diagnosed Hodgkin's disease: a prospective, multi-institutional AIDS clinical trials group study (ACTG 149). J Acquir Immune Defic Syndr. 2000 Aug 15;24(5):444-50. doi: 10.1097/00126334-200008150-00009. PMID 11035615
- [Background] Levine AM, et al. Prospective, multicenter phase II trial of ABVD chemotherapy with G-CSF in HIV-infected patients with Hodgkin's disease (HD): AIDS Clincial Trials Group (ACTG) Study 149. Proc Annu Meet Am Soc Clin Oncol. 1997;16:A194